CLINICAL TRIAL: NCT04045379
Title: LASER and Radiofrequency as Alternative Treatments for Genitourinary Syndrome of Menopause
Brief Title: LASER and Radiofrequency and Genitourinary Syndrome of Menopause
Acronym: EPMLARF-arm1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ana Maria Homem de Mello Bianchi, Principal investigador, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP0431/2018 arm 1
Record Dates: First submitted 2019-05-20; First posted 2019-08-05 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Postmenopausal Atrophic Vaginitis; Postmenopausal Symptoms; Genitourinary Symptoms
Keywords: postmenopause; atrophic vaginitis; vulvovaginal atrophy; treatment; LASER; Radiofrequency; estriol; strogen therapy
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Lasers; Lasers, Gas; Estriol

STUDY DESIGN:
Intervention Model Description: The patient will be randomized in block to receive one of the three intravaginal therapies: LASER, Radiofrequency and topic estriol
Who Masked: Outcomes Assessor
Masking Description: the outcomes assessor will not know which therapy was used by the patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LASER (Active Comparator): The patients will receive 3 consecutive applications of intravaginal and vulvar CO2 (carbon dioxide)LASER, according to the manufacturer protocol for vaginal atrophy. The applications will be separated by the interval of 30 days
  Interventions: Procedure: LASER
- Micro Ablative Radiofrequency (Active Comparator): The patients will receive 3 consecutive applications of intravaginal and vulvar MIcro ablative radiofrequency, according to the manufacturer protocol for vaginal atrophy. The applications will be separated by the interval of 30 days
  Interventions: Procedure: Microablative Radiofrequency
- Estriol (Active Comparator): The patient will use intravaginal estriol, daily for 2 weeks and them twice a week for 3 months . Each 30 days, the patients will have an appointment when will be checked the weight of the estriol tube to verify the correct use.
  Interventions: Drug: Estriol

INTERVENTIONS:
Procedure: LASER — Use of the SmartXide Touch V²LR, Co2 Laser System to perform ambulatory intravaginal and vulvar application of LASER, to postmenopausal genitourinary syndrome. The patient will be in gynecological position, after remove of vaginal secretion, with gauze and under topic anesthesia, the LASER will be applied, according to the protocol of the manufactured.
  Other Names: Fractional Co2 (carbon dioxide)Laser; MonaLisa Touch® treatment; SmartXide Touch V²LR® Deka
  Arms: LASER
Procedure: Microablative Radiofrequency — Use of Linly™ equipment to perform ambulatory intravaginal and vulvar application of fractionated microablative radiofrequency, to postmenopausal genitourinary syndrome. The patient will be in gynecological position, after remove of vaginal secretion, with gauze and under topic anesthesia, the radiofrequency will be applied, according to the protocol of the manufactured.
  Other Names: FRAAX; Linly™ Loktal Medical Electronics
  Arms: Micro Ablative Radiofrequency
Drug: Estriol — The patient will perform self application of this vaginal estriol daily for 2 weeks and after that the applications will occur twice a week.
  Other Names: Estriol 01mg/ml
  Arms: Estriol

SUMMARY:
This is a randomized controlled trial to evaluate the use of LASER, Micro Ablative radiofrequency and topic strogen to treat symptoms of vulvovaginal atrophy of post menopause.

DETAILED DESCRIPTION:
Post menopause women with moderate or severe signs or symptoms of vulvovaginal atrophy will be eligible for the study.

The patients will be randomized to receive one of the three intravaginal therapies: LASER, Micro Ablative radiofrequency or Estriol. The applications will occur in the interval of 30 days for 3 times, for LASER and Radiofrequency groups. For the estriol group, the application will be done by the patient, daily for 2 weeks and them twice a week for 3 months, and each 30 days, the patients will have an appointment when will be checked the weight of the estriol tube, to verify the correct use.

The follow-up visits will occur 30, 90, 180 and 360 days after the conclusion of the third month of treatment.

Will be evaluated: vulvar and vaginal histology before and after the use of LASER, radiofrequency or estriol; microbiota and vaginal pH before and after the use of LASER, radiofrequency or estriol; extracellular matrix and metalloproteinases in the remodeling of vulvovaginal collagen induced by estrogen, LASER and radiofrequency; quality of life, sexual dysfunctions and complaints before and after the use of LASER, radiofrequency or hormones; metabolomics and vaginal microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 2 and 5 years after menopause, without hormone therapy for at least 2 years
2. To present, at least moderate, or severe intensity (score 4 or more of visual analog scale ( 0-10)) of one of the signs or symptoms of of vulvovaginal atrophy:

   * Burning
   * Discomfort
   * Dryness
   * Cracks
   * Pruritus
   * Lack of vaginal lubrication
   * Penetration dyspareunia that began at the menopausal or postmenopausal transition
   * Decreased vaginal epithelium turgor and trophism
   * Deletion of mucous and skin folds.

The Exclusion criteria will be:

1. Active genital infection, active infection of HPV (human papillomavirus) or Herpes, users of medications with estrogenic effect (digoxin, tamoxifen and other chemicals)
2. Postmenopausal genital bleeding, uncontrolled diabetes, use of multivitamins with zinc, use of copper or hormonal IUDs (intrauterine device) at the time of inclusion, presence of genitourinary or rectovaginal fistulas.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Clinical Improvement of signs and symptoms postmenopausal genitourinary syndrome with intravaginal LASER, Microablative Radiofrequency, and topic estriol | The evaluation will be done 180 days after treatment
  Will be applied a Visual Analogic Scale (0-10) to access the improvement of genitourinary signs and symptoms, the results of the three groups will be compared
Satisfaction of postmenopausal women with genitourinary syndrome with the treatment by intravaginal LASER, Micro ablative Radiofrequency, and topic estriol | The evaluation will be done 180 days after treatment
  Will be applied a LIKERT Satisfaction Scale (1-5) to access the satisfaction with the treatment, the results of the three groups will be compared

SECONDARY OUTCOMES:
Evaluation of Microbiota before and after the use of intravaginal LASER, Micro Ablative radiofrequency or topic estriol. | The evaluation will occur pre treatment 30, 90 , 180 and 360 days after treatment
  The vaginal flora will be evaluated by vaginal smear. The results of the three groups will be compared
Evaluation of vaginal pH before and after the use of intravaginal LASER, Micro ablative radiofrequency or topic estriol. | The evaluation will occur pre treatment and 30, 90, 180 and 360 days after treatment
  The vaginal pH will be verified by the use of pH tape's .The results of the three groups will be compared
Histologic evaluation of vagina and vulva before and after the use of intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic estriol. | The evaluation will occur pre treatment and 30 days after treatment
  Thickness of epithelium (mm and number of layers), and evaluation of expression of Ki-67 and VEGF (vascular endothelial growth factor) will be done on vaginal and vulvar biopsies.The results of the three groups will be compared
Evaluation of impact in Quality of life after treatment with intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic estriol. | The evaluation will occur pre treatment and 30 days after treatment
  The IQol (incontinence quality of life questionnaire, validated to portuguese language - score 0-100) will be used to evaluate quality of life .The results of the three groups will be compared
Evaluation of impact in Sexual function after treatment with intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic estriol. | The evaluation will occur pre treatment and 30 days after treatment
  The FSF-I(Female Sexual Function Index , validated to portuguese language- score range from 2 - 36) will be used to evaluate sexual function . The results of the three groups will be compared
Evaluation of extracellular matrix before and after the use of intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic estriol. | The evaluation will occur pre treatment and 30 days after treatment
  Evaluation of the composition and concentration of the glycosaminoglycans of extracellular matrix in the vaginal and vulvar biopsies by specific markers. The results of the three groups will be compared
Evaluation of matrix metalloproteinases(MMP) in remodeling of vulvovaginal collagen induced by intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic estriol. | The evaluation will occur pre treatment and 30 days after treatment
  Evaluation of the tissue distribution of the MMP-1, MMP-2, MMP-3, MMP-7, MMP-9 metalloproteinases of collagen I, II, IV and elastin proteins by specific markers on vaginal and vulvar biopsies. The results of the three groups will be compared
Evaluation of visual aspect of vulva after the use of intravaginal and vulvar LASER, Micro Ablative radiofrequency or topic estriol. | The pictures will be taken before and 30 days and 180 days after treatment.
  Pictures of vulva will be taken before and after treatment. The images will be evaluated by a blind gynecologist and dermatologist regarding the type of treatment and the chronological order of the photos, which will classify the images as: better; equal or worse, in relation to tropism and number of vulvar skin grooves, The results of the three groups will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Zsuzsanna IK Jarmy - di Bella, PhD, Study Chair — Professor
Locations (1):
- Federal University of Sao Paulo - Unifesp, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Oliveira CD, de Mello Bianchi AMH, Campos MLP, Nogueira MCC, Sartori MGF, de Gois Speck NM. Women with Genitourinary Syndrome of Menopause Treated with Vaginal Estriol, Microablative Fractional CO2 Laser and Microablative Fractional Radiofrequency: A Randomized Pilot Study. Photobiomodul Photomed Laser Surg. 2023 Dec;41(12):718-724. doi: 10.1089/photob.2023.0113. PMID 38085184